CLINICAL TRIAL: NCT00370136
Title: Sentinel Node Diagnostics With Ultrasound Contrast in Melanoma
Brief Title: Sentinel Node With Ultrasound Contrast in Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: (KF)01288200
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Last update posted 2008-06-18 (Estimated); Status verified 2008-06

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Drug: ultrasound contrast

SUMMARY:
The purpose is to evaluate,in 20 patients, if the sentinel node(s) in melanoma can be detected by lymph contrast ultrasound. In comparing the patients will also get lymph-scintigraphy and sentinel node detection wiht blue dye.

The goal is to improve the method for detecting sentinel node(s) in melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Malignant melanoma on a extremity,
* No spread of the cancer,
* Patients over 18 years old,

Exclusion Criteria:

* Pregnancy,
* Lactating,
* Severe hart disease,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-03; Study Completion 2008-04

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Nielsen, MDSc, Principal Investigator — Department of Radiology, section ultrasound
Locations (1):
- Copenhagen univercity hospital, Department of Radiology, section of ultrasound, Copenhagen, Denmark